CLINICAL TRIAL: NCT03903640
Title: Phase II Study of Optune Device - TT Field Plus Nivolumab and Ipilimumab for Melanoma With Brain Metastasis
Brief Title: Optune Device - TT Field Plus Nivolumab and Ipilimumab for Melanoma With Brain Metastasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early on 03/09/2022 due to low accrual during the COVID-19 pandemic.
Sponsor: Washington University School of Medicine (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201903162
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Results first posted 2022-05-12 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Melanoma With Brain Metastasis
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Optune + Ipilimumab + Nivolumab (Experimental): * Ipilimumab at 3 mg/kg IV over 90 minutes on Day 1 of each 21-day cycle for 4 cycles.
  * Nivolumab at 1 mg/kg IV over 30 minutes on Day 1 of each 21-day cycle for 4 cycles, then at 240 mg IV over 30 minutes on Days 1 and 15 of each 28-day cycle for up to 20 doses
  * Within 2 weeks of the start of ipilimumab (before or after), treatment with Optune will begin. All patients will be required to shave their heads to initiate array placement and Optune therapy.
  * Treatment may continue for up to 1 year
  Interventions: Device: Optune; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Device: Optune — -Optune is programmed by Novocure to deliver 200 kHz TTFields in two sequential, perpendicular field directions at a maximal intensity of 707mARMS.
Biological: Nivolumab — -Standard of care
  Other Names: Opdivo
Biological: Ipilimumab — -Standard of care
  Other Names: Yervoy

SUMMARY:
This phase II study will evaluate the safety of combining intermediate frequency electric field (TT Field) with immunotherapy in melanoma patients with brain metastasis. The data of this study will also inform whether this combination will offer advantage in progression free survival (PFS) and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed melanoma with metastasis to the brain.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 10 mm with CT scan or MRI, as ≥ 20 mm by chest x-ray, or ≥ 10 mm with calipers by clinical exam.
* Candidate for treatment with immunotherapy.
* At least 18 years of age.
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation, including at least 5 months (for women of childbearing potential) and at least 7 months (for men) after last dose of study drug. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Received treatment in the metastatic setting
* Treated with whole brain radiation Receiving targeted therapy or on immunosuppressive agents (dexamethasone> 4mg/day) within 1 week of therapy.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, ipilimumab, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* History of pre-existing immunodeficiency disorder or autoimmune condition requiring immunosuppressive therapy. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines.
* Known sensitivity to conductive hydrogels.
* Skull defects such as missing bone or bullet fragments.
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, vagus nerve stimulator, and other implanted electronic devices in the brain or spinal cord.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with nivolumab and/or ipilimumab. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2021-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Ansstas, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to enrollment on 07/01/2019 and closed to enrollment on 03/09/2022.
Period: Overall Study
Arm/Group | Optune + Ipilimumab + Nivolumab
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 59 [49 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Intracranial Progression-free Survival
Description: * The PFS time will be calculated as the duration of time from the date of first dose of study treatment to the date of earliest intracranial progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Time Frame: At 6 months (up to 184 days)
Measure: Median (Full Range); unit: days
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
days | 99.5 [15 to 184]

2. Secondary Outcome: Overall Survival
Description: -Defined as the duration of time from the date of first dose of study treatment to death from any cause.
Time Frame: At 6 months (up to 184 days)
Measure: Median (Full Range); unit: days
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
days | 104.5 [25 to 184]

3. Secondary Outcome: Best Intracranial Response Rate
Description: * Defined as the percentage of patients with a confirmed intracranial complete or partial response
  * Using modified RANO criteria
Time Frame: Until disease progression or death whichever comes first (median follow-up 53 days (full range 15-91 days))
Measure: Count of Participants; unit: Participants
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
Participants | 0

4. Secondary Outcome: Best Extracranial Response Rate
Description: * Defined as the percentage of patients with a confirmed extracranial complete or partial response
  * Using modified RANO criteria
Time Frame: Until disease progression or death whichever comes first (median follow-up 53 days (full range 15-91 days))
Measure: Count of Participants; unit: Participants
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
Participants | 0

5. Secondary Outcome: Extracranial Progression-free Survival
Description: * Defined as the duration of time from the date of first dose of study treatment to the date of earliest extracranial progression or death, whichever occurs first. Patients who neither progress nor die by the data cutoff date will be censored at the last follow up.
  * Using modified RANO criteria
Time Frame: At 6 months
Measure: Median (Full Range); unit: days
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
days | 58 [25 to 91]

6. Secondary Outcome: Safety of the Treatment Regimen as Measured by Number of Participants With Treatment-related Grade 3 or Greater Adverse Events
Description: -The descriptions and grading scales found in CTCAE version 5.0.
Time Frame: Through 100 days after completion of treatment (median follow-up 107.5 days, full range (25 days-190 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
Participants | 0

7. Secondary Outcome: Safety of the Treatment Regimen as Measured by Number of Participants With Discontinuations Due to Treatment Related Adverse Events.
Description: -The descriptions and grading scales found in CTCAE version 5.0.
Time Frame: Through 100 days after completion of treatment (median follow-up 107.5 days, full range (25 days-190 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Optune + Ipilimumab + Nivolumab
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were followed from start of treatment until 100 days after last day of treatment (median follow-up 107.5 days, full range (25 days-190 days)). All-cause mortality was followed from time of enrollment until completion of follow-up (median follow-up 314.50 days (full range 25 days-604 days)
Arm/Group | Optune + Ipilimumab + Nivolumab
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optune + Ipilimumab + Nivolumab (N=2)
Death NOS (General disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Optune + Ipilimumab + Nivolumab (N=2)
Anemia (Blood and lymphatic system disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Metabolism and nutrition disorders) | 1
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Confusion (Psychiatric disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The study was opened to enrollment from 07/01/2019 through 03/09/2022. The study was terminated early due to low enrollment. The low enrollment was due to the COVID-19 pandemic and no external referrals for the trial. The Principal Investigator reached out to other academic institutions about opening the trial but there was not any interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT03903640/Prot_SAP_001.pdf